CLINICAL TRIAL: NCT03701009
Title: Saline Irrigation Reduces the Residual Bile Duct Stones After ERCP: a Single-arm Prospective Study
Brief Title: Saline Irrigation Reduces the Residual Bile Duct Stones During Endoscopic Retrograde Cholangiopancreatography (ERCP)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hepatopancreatobiliary Surgery Institute of Gansu Province (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Saline irrigation in ERCP
Record Dates: First submitted 2018-10-06; First posted 2018-10-09 (Actual); Last update posted 2020-07-14 (Actual); Status verified 2020-07

CONDITIONS: Stone Clearance
Keywords: ERCP; Common bile duct stone; Cholangitis; Residual stone; Irrigation
MeSH Terms: conditions — Gallstones; Cholangitis | interventions — Sodium Chloride

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Stone removal (Saline 50ml each time) (Other): After CBD stone removal via lithotripsy, and the cholangiogram showed normal, residual CBD stones were detected by SpyGlass in the first round, if CBD not clean, sterile saline 50ml were intermittently irrigated into the CBD. After that, if bile duct clearance was not achieved, another 50ml saline will be irrigated into CBD again until the clear bile duct determined by SpyGlass.
  Interventions: Procedure: CBD stone removal via lithotripsy; Procedure: Saline 50ml; Procedure: Saline +50ml

INTERVENTIONS:
Procedure: CBD stone removal via lithotripsy — Hold saline irrigation just after X-ray demonstrated no stone residue, a Spyglass explored.
Procedure: Saline 50ml — If not clean, intermittent saline irrigation 50ml, and Spyglass explored second time.
Procedure: Saline +50ml — If still have some stone fragments, intermittent saline irrigation another 50ml after the second Spyglass detection, Spyglass explored third time to evaluate stone clearance.

SUMMARY:
The purpose of this study was to evaluate the usefulness of saline solution irrigation in decreasing residual common bile duct (CBD) stones.

DETAILED DESCRIPTION:
In recent years, ERCP is the standard procedure to remove the bile duct stones. The big stones(>1.2 cm) require additional lithotripsy procedures for complete stone removal. Nevertheless, small stone fragments still remain in the common bile duct when the cholangiogram shows normal. The fragments are too small to be verified. These retained fragments may cause recurrence of stones. Another way to demonstrate residual CBD stones is to use intraductal ultrasonography (IDUS). However, IDUS has limited availability in clinical practice. The single-operator cholangioscopy (SOC)-system Spyglass gains widespread acceptance because of its independent washing channels and direct viewing. The investigators used Spyglass to detect if saline(50 or 100ml) infusion might clear the bile duct fragments after ERCP. Saline irrigation has many advantages such as easy stone removal, no additional cost and rare side effects. The purpose of this study is to evaluate the usefulness of saline solution irrigation in decreasing residual CBD stones.

ELIGIBILITY:
Inclusion Criteria:

* ERCP common bile duct stone patients were able to provide written informed consent;
* Size of stone large than 1.2 cm.

Exclusion Criteria:

* Unwillingness or inability to consent for the study;
* Coagulation dysfunction (INR> 1.5) and low peripheral blood platelet count (<50×10^9 / L) or using anti-coagulation drugs;
* Previous ERCP;
* Prior surgery of Bismuth Ⅱ, Roux-en-Y and Cholangiojejunostomy;
* Preoperative coexistent diseases: acute pancreatitis, GI tract hemorrhage or perforation, severe liver disease(such as decompensated liver cirrhosis, liver failure and so on), septic shock;
* Biliary-duodenal fistula confirmed during ERCP;
* Pregnant women or breastfeeding;
* Presence of intrahepatic duct stone;
* Malignancy.

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 47 (Actual)
Dates: Start 2018-10-10 (Actual); Primary Completion 2020-07-01 (Actual); Study Completion 2020-07-01 (Actual)

PRIMARY OUTCOMES:
Stone fragments clearance | 3 months
  Type 1: Not clean, large stone fragments; Type 2: Clusters residue and floccule; Type 3: Small biliary sludge or floccule Type 4: Slightly clean with a small amount of floccule or small residue; Type 5: Clean.

SECONDARY OUTCOMES:
Post-ERCP cholangitis | 3 months
  Number of Post-ERCP cholangitis participants, Post-ERCP cholangitis was defined as a temperature of more than 38 °C for 24-48 h after the procedure, thought to have a biliary cause without evidence of other concomitant infections.
Bleeding | 3 months
  Number of Bleeding participantsas who was defined as the clinical and endoscopic evidence of hemorrhage associated. with a decreasing the hemoglobin level >2 g/dl.
Post-ERCP pancreatitis | 3 months
  Number of Post-ERCP pancreatitis participants who was defined as any new or worsened abdominal pain with an increasing serum. amylase of over three times the upper normal limit that was measured more than 24h after the procedure.
Perforation | 3 months
  Number of perforation participants who was defined as the presence of air or contrast in the retroperitoneal space.
The procedure time | 3 months
  Was defined as the sum of times of all processes of endoscopic procedure.

CONTACTS AND LOCATIONS:
Overall Officials: Xun Li, MD,PhD, Study Director — Hepatopancreatobiliary Surgery Institute of Gansu Province
Locations (1):
- Hepatopancreatobiliary Surgery Institute of Gansu Province, Lanzhou, Gansu, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Ahn DW, Lee SH, Paik WH, Song BJ, Park JM, Kim J, Jeong JB, Hwang JH, Ryu JK, Kim YT. Effects of Saline Irrigation of the Bile Duct to Reduce the Rate of Residual Common Bile Duct Stones: A Multicenter, Prospective, Randomized Study. Am J Gastroenterol. 2018 Apr;113(4):548-555. doi: 10.1038/ajg.2018.21. Epub 2018 Mar 27. PMID 29610513
- [Background] Ramchandani M, Reddy DN, Gupta R, Lakhtakia S, Tandan M, Darisetty S, Sekaran A, Rao GV. Role of single-operator peroral cholangioscopy in the diagnosis of indeterminate biliary lesions: a single-center, prospective study. Gastrointest Endosc. 2011 Sep;74(3):511-9. doi: 10.1016/j.gie.2011.04.034. Epub 2011 Jul 7. PMID 21737076